CLINICAL TRIAL: NCT00901342
Title: An Open Label Study of Sipuleucel-T in Men With Metastatic Castrate Resistant Prostate Cancer
Brief Title: Open Label Study of Sipuleucel-T in Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P09-1
Record Dates: First submitted 2009-05-07; First posted 2009-05-13 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: Androgen independent prostate cancer (AIPC); CRPC; prostate cancer; prostate; immune therapy; immunotherapy; vaccine; dendritic cells; antigen-presenting cells; antigen presenting cells; cancer vaccine; prostate specific antigen (PSA); prostatic adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sipuleucel-T (Experimental): Subjects received infusion of sipuleucel-T, at 2-week intervals, for a total of 3 infusions.
  Interventions: Biological: sipuleucel-T

INTERVENTIONS:
Biological: sipuleucel-T — Sipuleucel-T is an autologous cellular product consisting of antigen presenting cells (APCs) activated with PA2024, a recombinant fusion protein composed of prostatic acid phosphatase (PAP), linked to granulocyte-macrophage colony-stimulating factor (GM-CSF)
  Other Names: • Provenge® • APC8015

SUMMARY:
This is a Multicenter, Open Label, Phase 2 Study of Sipuleucel-T in Men with Metastatic Castrate Resistant Prostate Cancer (CRPC).

DETAILED DESCRIPTION:
Subjects received sipuleucel-T at 2-week intervals, for a total of 3 infusions. The study evaluated the safety and magnitude of the immune responses to treatment with sipuleucel-T. All subjects were followed for 30 days following the last infusion of sipuleucel-T. Following the Study Completion Visit, survival, treatment-related serious adverse event (SAE)s and cerebrovascular event (CVE)s were collected via Long Term Follow-up Telephone Assessment occurring Q6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the prostate
* Metastatic disease
* Castrate resistant prostate cancer
* Castrate level of testosterone (< 50 ng/dL) achieved via medical or surgical castration
* Life expectancy of ≥ 3 months
* Men ≥ 18 years of age
* Adequate hematologic, renal and liver function

Exclusion Criteria:

* Presence of known lung, liver, or brain metastases
* Evidence of neuroendocrine or small cell features
* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* Prior treatment with 3 infusions of sipuleucel-T (infusions of APC8015F are not exclusionary)
* Imminent pathologic long-bone fracture (cortical erosion on radiography > 50%) or spinal cord compression
* Known malignancies other than prostate cancer that are likely to require treatment within six months of registration
* A requirement for systemic immunosuppressive therapy for any reason
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to Sipuleucel-T or granulocyte-macrophage colony-stimulating factor
* Any infection requiring parenteral antibiotic therapy or causing fever (temp > 100.5F or > 38.1C) within 1 week prior to registration
* Any medical intervention or other condition which, in the opinion of the Principal Investigator or the Dendreon Medical Monitor, could compromise adherence with study requirements or otherwise compromise the study's objectives

Treatment with any of the following medications or interventions within 28 days of registration:

* Systemic corticosteroids. Use of inhaled, intranasal, intra-articular, and topical steroids is acceptable, as is a short course (ie, ≤ 1 day) of corticosteroids to prevent a reaction to the IV contrast used for CT scans
* Non-steroidal anti-androgens (eg, bicalutamide, flutamide, or nilutamide)
* External beam radiation therapy or major surgery requiring general anesthetic
* Any other systemic therapy for prostate cancer including secondary hormonal therapies, such as megestrol acetate (Megace®), diethylstilbestrol (DES), and ketoconazole. Medical castration therapy is not exclusionary
* Chemotherapy
* Treatment with any other investigational product

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-10; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Israel, MD, Study Director — Valeant Pharmaceuticals North America LLC
Locations (18):
- United States (18):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - The University of Chicago Medical Center, Chicago, Illinois
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Indiana University Department of Urology, Indianapolis, Indiana
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - Hematology Oncology Consultants, Greenbelt, Maryland
  - Myron I. Murdock MD LLC, Greenbelt, Maryland
  - John Theurer Cancer Center at Hackensack, Hackensack, New Jersey
  - NYU Cancer Institute, New York, New York
  - Mount Sinai School of Medicine Department of Urology, New York, New York
  - Columbia University Medical Center, New York, New York
  - GU Oncology Research Program, Durham, North Carolina
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology, PA - Sammons Cancer Center, Dallas, Texas
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
  - Virginia Mason Medical Center Urology and Renal Transplantation, Seattle, Washington
  - Aurora Advanced Healthcare, Inc, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: US TOO International — http://www.ustoo.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sipuleucel-T
Started | 104
Received at Least 1 Infusion | 98
Completed | 89 (89 subjects completed the study completion visit)
Not Completed | 15
Not completed — Adverse Event | 1
Not completed — Death | 4
Not completed — Disease progression | 1
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 73
Age, Continuous [Mean (Full Range); unit: years] | 69.2 [46.0 to 91.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 104
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 4
  White | 95
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 104
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — ECOG Performance Status is a method used to assess the functional status of a patient. The scale ranges from 0-5. 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out light or sedentary work; 2=Ambulatory, capable of all self-care but unable to carry out work activities. Up and about >50% of waking hour; 3=Capable of limited self-care, confined to bed or chair >50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead
  Participants
    ECOG 0=Fully Active; No restrictions. | 66
    ECOG 1= Restricted Strenuous Activity | 35
    ECOG 2=Ambulatory, capable of self-care; no work | 3
Gleason Score [Count of Participants; unit: Participants] — Gleason score= prostate cancer grading system based on how tissue looks under a microscope. Scores range 2-10 and indicates how likely it is that a tumor will spread. A low score means the cancer tissue is similar to normal tissue and the tumor is less likely to spread. Gleason Score ≤ 6=the tumor is well differentiated, less aggressive and likely to grow more slowly;7=the tumor is moderately differentiated, moderately aggressive, and likely to grow but may not spread quickly;≥8=the tumor is poorly differentiated or undifferentiated, highly aggressive, and likely to grow faster and spread.
  Participants
    Gleason Score ≤ 6 | 16
    Gleason Score = 7 | 35
    Gleason Score ≥ 8 | 51
    Gleason Score Missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received At Least 1 Infusion of Sipuleucel-T in Men With Metastatic Castrate-resistant Prostate Cancer (CRPC)
Time Frame: Day 0 (first infusion) and up to 3 infusions at 2-week intervals
Population: Participants who Received At least 1 Infusion
Measure: Number; unit: participants
Groups:
- Sipuleucel-T: All subjects who received ≥ one sipuleucel-T infusion
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 98
participants | 98

ADVERSE EVENTS:
Time Frame: Subjects were assessed for safety not less than 30 days post-final infusion with sipuleucel-T. Following the Study Completion Visit, survival, treatment-related serious adverse events, and cerebrovascular events (CVE)s were collected via Long Term Follow-up Telephone Assessment every 6 months until subject death or study conclusion.
Description: Adverse events were reported in the safety population. The safety population consisted of all subjects who underwent at least 1 infusion.
Arm/Group | Sipuleucel-T
All-Cause Mortality (participants affected / at risk) | 4/98
Serious Adverse Events (participants affected / at risk) | 13/98
Other Adverse Events (participants affected / at risk) | 91/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T (N=98)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T (N=98)
Anaemia (Blood and lymphatic system disorders) | 6 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Dizziness (Nervous system disorders) | 9 (10)
Headache (Nervous system disorders) | 8 (11)
Anxiety (Psychiatric disorders) | 7 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Asthenia (General disorders) | 6 (6)
Citrate toxicity (Injury, poisoning and procedural complications) | 6 (8)
Hypertension (Vascular disorders) | 6 (7)
Oedema peripheral (General disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 6 (6)
Contusion (Injury, poisoning and procedural complications) | 5 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7)
Fatigue (General disorders) | 28 (35)
Nausea (Gastrointestinal disorders) | 18 (21)
Chills (General disorders) | 17 (25)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11)
Paraesthesia oral (Gastrointestinal disorders) | 11 (18)
Constipation (Gastrointestinal disorders) | 10 (10)
Pyrexia (General disorders) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study will be published and/or presented in an integrated manner reflecting the results observed across all participating centers. Accordingly, decisions on timing and content of publications and presentations relating to the Study will be coordinated by Dendreon in communication with institutions contributing patients to the Study.